CLINICAL TRIAL: NCT03912350
Title: The Effect of Hepatic Impairment on the Pharmacokinetics of Balovaptan: A Phase I, Multiple-Center, Open-Label Study Following Multiple Daily Oral Doses of Balovaptan in Subjects With Moderate Hepatic Impairment and Healthy Subjects With Normal Hepatic Function
Brief Title: The Effect of Hepatic Impairment on the Pharmacokinetics of Balovaptan
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is on hold due to stopping of the Autism Spectrum Disorder program with balovatpan, the study drug.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP41045
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — balovaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Participants with moderate hepatic impairment.
  Interventions: Drug: Balovaptan
- Reference group (Active Comparator): Healthy pariticipants with normal hepatic function.
  Interventions: Drug: Balovaptan

INTERVENTIONS:
Drug: Balovaptan — Participants will receive 1 tablet of balovaptan once daily (QD) on Days 1 through 14.

SUMMARY:
This is a multi-center, non-randomized, open-label, parallel group, multiple-dose study to assess the pharmacokinetic, safety, and tolerability of balovaptan in male and female subjects with moderate hepatic impairment compared to healthy subjects with normal hepatic function matched by age (±10 years), sex, and body mass index (BMI; ±20%).

ELIGIBILITY:
Inclusion Criteria for All Participants:

* BMI between 18 and 40 kg/m2, inclusive.
* Women of childbearing potential must either: agree to use one highly effective contraceptive method combined with a barrier method from Screening until 90 days after the last dose of study drug or practice true abstinence because of the subject's lifestyle choice; be in an exclusively same-sex relationship.
* For men: agreement to use contraceptive measures
* Females of child-bearing potential must refrain from donating ova from Day -1 until 90 days after the safety Follow-up visit. Males must refrain from donating sperm from Day -1 until 90 days after the safety Follow-up visit.

Inclusion Criteria for Participants with Hepatic Impairment:

* Stable, documented moderate liver disease diagnosed >6 months and stable for at least 3 months prior to Screening.
* Participants with moderate hepatic impairment may have medical findings consistent with their hepatic dysfunction. Participants with abnormal findings considered in line with underlying hepatic disease by the Investigator will be eligible.

Inclusion Criteria for Healthy Participants:

* Healthy status is defined by no clinically significant findings from medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, chemistry, and urinalysis at Screening and/or Day -1 as assessed by the Investigator (or designee). Gilbert's syndrome is acceptable.

Exclusion Criteria for All Participants:

* History of significant hypersensitivity, intolerance, or allergy to any drug compound, constituents or excipients of the study drug, food, or other substance, unless approved by the Investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
* Evidence of hepatorenal syndrome and estimated creatinine clearance range <60 mL/min or abnormal and clinically significant sodium and potassium levels, as determined by the Investigator (or designee).
* Female subjects of childbearing potential with a positive serum pregnancy test at Screening and/or at admission (Day -1), or who are lactating.
* History of drug/chemical abuse within 2 years prior to Screening; current active substance abuse will not be permitted.
* Known personal or family history of congenital long QT syndrome or sudden unexplained death.

Exclusion Criteria for Participants with Hepatic Impairment:

* History within 3 months prior to Screening, or current symptoms of, hepatic encephalopathy Grade 2 and above.
* Evidence of severe ascites.
* Recent history of, or the treatment of, esophageal bleeding within 3 months of first dose, unless banded.
* Participants who have had a porto-systemic shunt.
* Participants who have a history of paracentesis within 3 months prior to Day -1.
* Participants who have a history of unstable diabetes mellitus as evidenced by hemoglobin A1c ≥ 9% at Screening.
* History of alcoholism within 3 months prior to Screening.
* Use of any prescription drugs within 30 days (or within 5 times the elimination half-life, if known, of the medication, whichever is longer) of first dose, with the exception of therapies for hepatic-associated disorders that have been stable for at least 60 days prior to first dose.
* Biliary liver cirrhosis or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Positive result on human immunodeficiency virus (HIV) 1, HIV2, Hepatitis B Surface Antigen (HBsAg).

Exclusion Criteria for Healthy Participants:

* History of presence of liver disease, injury, or dysfunction as indicated by any clinically significant deviations from normal reference ranges in liver function tests, unless approved by the Investigator of designee.
* Participants likely to need prescription medication during the study. Participants who have received any prescribed systemic or topical medication within 30 days (or within 5 times the elimination half-life, if known, of the medication, whichever is longer) of the first dose administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* Any slow-release medicinal formulations considered to still be active within 4 weeks (or within 5 times the elimination half-life of the medication, whichever is longer) prior to the first study drug administration are prohibited, unless in the opinion of the Investigator or designee the medication will not interfere with the study procedures or compromise safety.
* History of alcoholism within 2 years prior to Screening.
* Positive result on HIV 1, HIV2, HBsAg, Hepatitis B core antibody (HBcAb), and/or HCV antibody.
* Signs and symptoms potentially indicative of peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-26 (Estimated); Primary Completion 2022-09-24 (Estimated); Study Completion 2022-10-13 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of balovaptan | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16 hours post-dose on Day 1; pre-dose on Day 2 to Day 13; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Plasma concentration of M2 metabolite, as applicable | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16 hours post-dose on Day 1; pre-dose on Day 2 to Day 13; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Plasma concentration of M3 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16 hours post-dose on Day 1; pre-dose on Day 2 to Day 13; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
AUC during the dosing interval on Day 1 of balovaptan | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1
AUC during the dosing interval on Day 1 of M2 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1
AUC during the dosing interval on Day 1 of M3 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1
AUC during the dosing interval at steady state on Day 14 of balovaptan | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
AUC during the dosing interval at steady state on Day 14 of M2 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
AUC during the dosing interval at steady state on Day 14 of M3 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Maximum observed plasma concentration (Cmax) of balovaptan | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Maximum observed plasma concentration (Cmax) of M2 metabolite | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Maximum observed plasma concentration (Cmax) of M3 metabolite | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Time of maximum observed plasma concentration (Tmax) of balovaptan | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Time of maximum observed plasma concentration (Tmax) of M2 metabolite | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Time of maximum observed plasma concentration (Tmax) of M3 metabolite | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Metabolite:Parent ratio of area under the plasma (MRauc) of M2 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Metabolite:Parent ratio of area under the plasma (MRauc) of M3 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Metabolite:Parent ratio of maximum observed plasma (MRcmax) of M2 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Metabolite:Parent ratio of maximum observed plasma (MRcmax) of M3 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent volume of distribution (V/F) of balovaptan | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent volume of distribution (V/F) of M2 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent volume of distribution (V/F) of M3 metabolite | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Terminal phase rate constant (λZ) of balovaptan, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Terminal phase rate constant (λZ) of M2 metabolite, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Terminal phase rate constant (λZ) of M3 metabolite, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent terminal elimination half-life (t½) of balovaptan, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent terminal elimination half-life (t½) of M2 metabolite, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent terminal elimination half-life (t½) of M3 metabolite, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent plasma clearance after oral administration (CLss/F) of balovaptan, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent plasma clearance after oral administration (CLss/F) of M2 metabolite, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent plasma clearance after oral administration (CLss/F) of M3 metabolite, when possible | Pre-dose, and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent volume of distribution based on the terminal phase after oral administration (Vz/F) of balovaptan, when possible | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent volume of distribution based on the terminal phase after oral administration (Vz/F) of M2 metabolite, when possible | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14
Apparent volume of distribution based on the terminal phase after oral administration (Vz/F) of M3 metabolite, when possible | 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 1; pre-dose and 1, 2, 3, 4, 5, 6, 9, 12, 16, and 24 hours post-dose on Day 14

SECONDARY OUTCOMES:
Percentage of participants with adverse events | Up to approximately 18 weeks from screening (screening is up to 28 days prior to admission to the clinical research unit).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).